CLINICAL TRIAL: NCT03154762
Title: National Institute of Respiratory Diseases Mexico
Brief Title: Anti-inflammatory Effect of Nocturnal NIPPV on Acute Asthma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of Respiratory Diseases, Mexico (Other Government)
Responsible Party: Principal Investigator, Jose Luis Carrillo Alduenda, MD, National Institute of Respiratory Diseases, Mexico
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: C34-14
Record Dates: First submitted 2017-05-11; First posted 2017-05-16 (Actual); Last update posted 2019-08-28 (Actual); Status verified 2019-08

CONDITIONS: Asthma Acute
MeSH Terms: interventions — Continuous Positive Airway Pressure

STUDY DESIGN:
Intervention Model Description: Experimental, prospective, longitudinal, comparative, parallel group study
Who Masked: Participant, Investigator
Masking Description: Similar equipment will be used, the programming of the positive pressure device will be performed by an external person and a cover will be placed on the screen.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- NIPPV (Experimental): Patients will receive NIPPV with an S bilevel device during 4 nights, the equipment will be placed ad libitum, a 12 cmH2O inspiratory pressure and a 4 cmH2O expiratory pressure will be administered through a nasal mask. CRP, FEV1, exhaled fraction of nitric oxide, IL-4, IL-5, IL-13, IL-17, IgE, cell count will be measured before and after intervention.
  Interventions: Device: NIPPV
- CPAP (Sham Comparator): Patients will receive a 4 cmH2O continuous positive airway pressure device during 4 nights; this is the minimum pressure necessary to avoid death space with no effect on minute ventilation. The equipment will be placed ad libitum. Pressure will be administered through a nasal mask. CRP, FEV1, exhaled fraction of nitric oxide, IL-4, IL-5, IL-13, IL-17, IgE, cell count will be measured before and after sham intervention.
  Interventions: Device: CPAP

INTERVENTIONS:
Device: NIPPV — Application of chronic distension of the airway through NIPPV to produce a reduction in bronchial hyperreactivity.
  Other Names: bilevel
  Arms: NIPPV
Device: CPAP — 4 cmH2O CPAP as the minimum pressure necessary to mobilize the air flow and avoid the space death with no effect on the ventilation.
  Arms: CPAP

SUMMARY:
INTRODUCTION: Asthma is a disease characterized by inflammation of the airway and secondary contraction of smooth muscle. Treatment for the crisis consist in the use of local and / or systemic bronchodilators and anti-inflammatories, and it has been shown that mechanical ventilation to the airway through non-invasive positive pressure ventilation (NIPPV) decreases bronchial hyperreactivity and contractility of smooth muscle.

OBJECTIVES: To assess the effect of nocturnal NIPPV on local inflammation, systemic inflammation and the state of hypersensitivity in patients with asthma attack.

MATERIALS AND METHODS: We will include patients with severe asthma attacks requiring hospitalization, without indication for acute NIPPV, and will be randomized to receive NIPPV with an spontaneous (S) bilevel or continuous positive airway pressure (CPAP, control group), all patients will receive standard treatment; gasometric exchange, local inflammation (FEV1 and Exhaled fraction of nitric oxide), systemic inflammation (C reactive protein, IL-4, IL-5, IL-13 and IL-17 in peripheral blood) and the hypersensitivity state (eosinophilia and IgE) between both groups will be compared after 4 days of treatment.

DETAILED DESCRIPTION:
RESEARCH QUESTION What is the effect of non invasive positive pressure ventilation (NIPPV) on systemic inflammation in patients with asthma attacks?

JUSTIFICATION Asthma is a global public health problem and one of the primary causes of care at the National Institute of Respiratory Diseases in Mexico; when presented as a crisis is a serious condition that puts the life of the patient at risk; in vitro and in vivo studies have shown that the application of chronic airway distention using non-invasive mechanical ventilation produces a reduction in bronchial hyperreactivity in patients with asthma and may have a positive effect on the treatment of this condition independent of its effects on ventilation in the presence of acute respiratory failure.

HYPOTHESIS The use of NIPPV will improve systemic inflammation assessed by C reactive protein (CRP) in patients with severe asthmatic crisis.

OBJECTIVES

Main Objective:

To assess the effect of NIPPV on systemic inflammation measure through C reactive protein in acute asthma

Secondary objectives:

1. - To assess the effect of NIPPV on the days of hospital stay in patients with asthma attacks.
2. - To evaluate adherence to NIPPV in patients with asthma attacks.
3. - To evaluate the effect of NIPPV on PaO2, PaCO2 and SpO2 in patients with asthma attacks.
4. - To evaluate the effect of NIPPV on FEV1 and Exhaled fraction of nitric oxide in patients with asthma attacks.
5. - To evaluate the effect of NIPPV on serum levels of interleukin (IL)-4, IL-5, IL-13 and IL-17 in patients with asthma attacks.
6. - To assess the effect of NIPPV on total eosinophil count and Immunoglobulin (Ig) E level in patients with asthma attacks.

MATERIALS AND METHODS

1. Design: A prospective, longitudinal, comparative, parallel group study will be conducted; it was approved by the Science and Bioethics Committees of the National Institute of Respiratory Diseases Mexico with the code C34-14. In all cases, informed consent will be requested.
2. Place: It will be carried out in the emergency and hospitalization service of the National Institute of Respiratory Diseases "Ismael Cosío Villegas" at Mexico city.
3. - Procedures:

   * Clinical history.
   * Chest X-ray.
   * Berlin Questionnaire. The Berlin questionnaire is a self-administered questionnaire validated in Spanish to establish the risk of obstructive sleep apnea.
   * Arterial gasometry.
   * Blood cell count.
   * Ultrasensitive C-reactive protein.
   * Determination of IgE.
   * Spirometry and Exhaled fraction of nitric oxide according to international guidelines.
4. - Intervention: Patients included will be randomized to receive, 4 nights of noninvasive nocturnal positive pressure ventilation with an S Bilevel device with a 12 cmH2O inspiratory pressure and a 4 cmH2O expiratory pressure or a 4 cmH2O Continuous Positive Airway Pressure (CPAP), as a control group.

   The equipment will be placed at night ad libitum and retired the following day in the morning, in all cases a VPAP ST S8 RESMED will be used. If the patient needs to increase inspired oxygen fraction it will be performed with nasal tips during the day and a distal oxygen connector at night. In all cases a nasal mask will be used.

   Blood gasometry, blood cell count, CRP, serum IL-4, IL-5, IL-13, IL-17 and IgE, Spirometry and Exhaled fraction of nitric oxide will be repeated at day 4.
5. - Data Analysis A convenience sample of 20 patients was established. A balanced randomization will be performed. The variables were summarized according to their type and distribution. The comparison of dichotomous variables will be performed using Fisher's Exact test. The comparison of independent continuous variables will be carried out with U of Mann Whitney and the related variables will be analyzed with Wilcoxon Related Ranks Test.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of asthma, performed by a physician, with spirometry and stable treatment for at least 3 previous months.
* Severe asthma crisis and hospitalization requirement of at least 4 days.

Exclusion Criteria:

* Life-threatening crisis.
* Requirement of Invasive or Non-Invasive Mechanical Ventilation.
* High risk for Obstructive Sleep Apnea (measured through the Berlin questionnaire).
* Active smoking.
* Another chronic lung disease other than asthma.
* Pneumonia (defined by the presence of an opacity of the lung parenchyma on a chest x-ray).
* Ischemic heart disease.
* Uncontrolled systemic arterial hypertension.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2017-10-31 (Actual); Study Completion 2017-10-31 (Actual)

PRIMARY OUTCOMES:
Systemic Inflammation | 4 days
  To evaluate the effect of NIPPV on C reactive protein in patients with asthma attacks.

SECONDARY OUTCOMES:
Hospitalization | 4 days
  To evaluate the effect of NIPPV on the days of hospital stay in patients with asthma attacks.
Adherence | 4 days
  To evaluate adherence to NIPPV in patients with asthma attacks
Gas Exchange | 4 days
  To evaluate the effect of NIPPV on PaCO2, PaO2 and SaO2 in patients with asthma attacks.
Local Inflammation | 4 days
  To evaluate the effect of NIPPV on FEV1 and exhaled fraction of nitric oxide in patients with asthma attacks.
Serum Inflammation | 4 days.
  To evaluate the effect of NIPPV on serum IL-4, IL-5, IL-13 e IL-17 in patients with asthma.attacks.

CONTACTS AND LOCATIONS:
Overall Officials: Jose Luis Carrillo Alduenda, Principal Investigator — Instituto Nacional de Enfermedades Respiratorias
Locations (1):
- Instituto Nacional de Enfermedades Respiratorias, Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: Yes
Through this organization and will be provided at the individual request of each interested researcher.

REFERENCES:
- [Result] Lafond C, Series F, Lemiere C. Impact of CPAP on asthmatic patients with obstructive sleep apnoea. Eur Respir J. 2007 Feb;29(2):307-11. doi: 10.1183/09031936.00059706. Epub 2006 Oct 18. PMID 17050561
- [Result] Xue Z, Yu Y, Gao H, Gunst SJ, Tepper RS. Chronic continuous positive airway pressure (CPAP) reduces airway reactivity in vivo in an allergen-induced rabbit model of asthma. J Appl Physiol (1985). 2011 Aug;111(2):353-7. doi: 10.1152/japplphysiol.01345.2010. Epub 2011 Apr 14. PMID 21493723
- [Result] Salerno FG, Pellegrino R, Trocchio G, Spanevello A, Brusasco V, Crimi E. Attenuation of induced bronchoconstriction in healthy subjects: effects of breathing depth. J Appl Physiol (1985). 2005 Mar;98(3):817-21. doi: 10.1152/japplphysiol.00763.2004. Epub 2004 Oct 8. PMID 15475599